CLINICAL TRIAL: NCT07045298
Title: Real-Time Continuous Glucose Monitoring for the Management of Patients With Type 2 Diabetes and Acutely Decompensated Heart Failure
Brief Title: CGM Use in Heart Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: American Heart Association (Other); Abbott Diabetes Care (Industry)
Responsible Party: Principal Investigator, Kasra Moazzami, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00007814; 2025P009798 (Other: Emory IRB)
Record Dates: First submitted 2025-05-27; First posted 2025-07-01 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; Diabetes Mellitus
Keywords: Continuous Glucose Monitoring (CGM) system; Acute Decompensated Heart failure; Glycemic control; Inpatient; Bedside point-of-care capillary glucose monitoring
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- POC glucose meter with Blinded CGM (Control/standard of care) (Active Comparator): Participants in the standard-of-care study arm will be provided with a Bluetooth-enabled blood glucose (BG) meter and testing supplies. A blood glucose monitoring account will be established and linked to the research site. Participants will be asked to perform glucose testing from 1- 3x daily. Testing would involve a minimum of once-daily tests that should include random fasting and post-prandial measurements. All participants will also be wearing blinded CGM devices. Providers will adjust oral agents or insulin doses based on POC results.
  Interventions: Diagnostic Test: POC BG + Blinded CGM
- Real Time CGM (RT-CGM) (Experimental): Participants in the CGM group will wear a Libre 2 rt-CGM with hypoglycemia and hyperglycemia alarms, and providers will adjust insulin therapy based on CGM profile information. All participants will be instructed on CGM placement and care. Diabetes educators will provide training sessions in the CGM system. The diabetes educator will educate subjects on how the CGM system differs from the traditional blood glucose (BG) meter
  Interventions: Device: Libre 2 rt-CGM

INTERVENTIONS:
Device: Libre 2 rt-CGM — Freestyle Libre 2 consists of a sensor applied to the back of the upper arm. The sensor is a penny-sized flexible filament placed beneath the skin's surface to measure interstitial fluid. This sensor is applied utilizing a sensor applicator provided in the packaging. The sensor continuously reads interstitial glucose readings every minute and syncs with the Freestyle View app. The hypoglycemia alarm will be set to < 80 mg/dl (for prevention of low blood glucose levels). Participants will be instructed to provide 15 grams of carbohydrates in response to a hypoglycemia alarm. The hyperglycemia alarm will be set at 300 mg/dl. Participants will call the research team if they experience repeated episodes > 300 mg/dl (more than 2 episodes in a single day or 2 or more episodes in consecutive days). The research team will instruct the participant to check with their physician for a possible new insulin regimen, but they will be allowed to remain in the study.
  Other Names: FreeStyle Libre Pro Glucose Monitoring System; Continuous Glucose Monitoring (CGM) device
  Arms: Real Time CGM (RT-CGM)
Diagnostic Test: POC BG + Blinded CGM — Standard of care point-of-care (POC) capillary blood glucose (BG) monitoring will be done before meals and bedtime daily during the study participation for up to 3 months.
  Other Names: Standard of care capillary glucose test and blinded CGM
  Arms: POC glucose meter with Blinded CGM (Control/standard of care)

SUMMARY:
Heart failure (HF) is a major cause of hospital admissions in the US, with over 6 million hospital days annually.

More than 40% of hospitalized patients with HF have diabetes mellitus (DM), which increases the risk of recurrent hospitalizations for HF with reduced and preserved ejection fraction by more than two-fold. Current methods for assessing glycemic control do not consider fluctuations in blood glucose levels, known as glycemic variability. High glycemic variability is a poor prognostic marker for HF re-hospitalizations. Given the significant prevalence and impact of DM in individuals with HF, it is crucial to examine whether improving glycemic control and avoiding hypoglycemia could lead to a decrease in HF readmissions. Real-time continuous glucose monitoring (rt-CGM), which provides glucose measurements as frequently as every 5 minutes, has improved glycemic control in insulin-treated adults with DM compared to the standard of care, capillary point-of-care blood glucose testing (POC). Researchers will monitor participants during their hospital stay and 3 months after discharge.

DETAILED DESCRIPTION:
HF is one of the leading causes of hospitalization among older adults. Nearly 1 in 4 HF patients are readmitted within 30 days of discharge and despite various strategies, the re-hospitalization rates remain high. HF hospitalization has an impact on morbidity, mortality, and healthcare costs. Therefore, it is crucial to identify and implement effective strategies to reduce the health and economic burden of HF re-hospitalization. Diabetes mellitus (DM) is one of the most common comorbidities in HF, impacting approximately a third of all patients. Several studies have reported that HF patients with DM have higher rates of recurrent HF hospitalizations, longer durations of hospital stay, and significantly higher mortality compared to HF patients without DM. Given the high prevalence and impact of DM on HF prognosis, it is important to understand how optimizing DM control can affect and improve the prognosis in this population. Glucose monitoring is central to safe and effective management for individuals with DM, particularly those using insulin. Recent studies have shown that real-time (rt) continuous glucose monitoring (CGM), by providing glucose measurements as often as every 5 minutes, low and high glucose alerts, and glucose trend information, with the potential to better inform diabetes management decisions compared with episodic self-monitoring with a blood glucose meter.

This pilot study will examine the potential benefits of remote glucose monitoring by rt-CGM-driven decisions for the hospital and post-discharge management patients with comorbid HF and DM.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 90 years admitted with a diagnosis of acute decompensated heart failure (ADHF), New York Heart Association (NYHA) class II, III, or IV symptoms (Aim 1) and discharged with a clinical diagnosis of ADHF (Aim 2).
* Patients with diabetes treated with diet alone or oral antidiabetic agents, Glucagon-like peptide-1 receptor agonists (GLP1-RAs), or insulin after discharge

Exclusion Criteria:

* Age < 18 or > 90 years;
* Patients with a history of type 1 diabetes;
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study;
* Patients on ventricular assist devices;
* History of a heart transplant or listed for a heart transplant;
* History of cardiac surgery (within 90 days before enrollment) or planned cardiac interventions within the following 6 months;
* Female participants who are pregnant or breastfeeding at the time of enrollment into the study;
* Hospice care or expected life expectancy of less than 6 months;
* Patients who are expected to require Magnetic Resonance Imaging (MRI) procedures during hospitalization or after discharge.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Mean Daily BG concentration after discharge (DC) | After hospital discharge up to 12 weeks
  Glucose levels measured by RT-CGM compared to traditional glucose monitoring testing (POCT-BG)
Frequency of clinically significant hypoglycemia after discharge | After hospital discharge up to 12 weeks
  The mean number of clinically significant hypoglycemia (BG < 54 mg/dL (<3.0 mmol/L)) events. Measurements by the POCT glucose monitoring testing (control) and real-time CGM (rt-CGM).
Frequency of overall and nocturnal hypoglycemia events after discharge | After hospital discharge up to 12 weeks
  The mean number of events of nocturnal hypoglycemia per participant by control (blinded CGM) and real time CGM group. Nocturnal hypoglycemia occurs between 12:00 midnight and 6:00 ante meridiem (AM). Hypoglycemia is defined as BG < 70 mg/dL (<3.9 mmol/L) and clinically significant hypoglycemia is defined as BG < 54 mg/dL (<3.0 mmol/L).
Percentage of glucose readings and time within target of 70 - 180 mg/dl | After hospital discharge up to 12 weeks
  Glycemic control will be measured by the percent of BG readings: 70-180 mg/dL measured by the control (blinded CGM) and rt-CGM.
Percentage of time within target of 70 - 180 mg/dl | After hospital discharge up to 12 weeks
  Glycemic control will be measured by the percentage of time with BG: 70-180 mg/dL measured by the control (blinded CGM) and real-time CGM
Frequency of hyperglycemia > 180 mg/dl and >250 mg/dl | After hospital discharge up to 12 weeks
  Number of events with hyperglycemia, defined as BG between 181 mg/dl and 249 mg/dl by traditional glucose monitoring testing (control) and real-time CGM group.
Percent of time with hyperglycemia | After hospital discharge up to 12 weeks
  Glycemic control will be measured by the percentage of the time with hyperglycemia > 180 mg/dl and > 250 mg/dl by traditional glucose monitoring testing (control) and by CGM (real-time)
Glycemic variability | After hospital discharge up to 12 weeks
  Glycemic variability will be calculated by glucose values obtained from the control (blinded CGM) and rt-CGM devices using standard deviation and coefficient of variation. It is designed to assess major glucose swings and exclude minor ones

SECONDARY OUTCOMES:
Composite number of HF re-hospitalization, emergency department/urgent clinic visits for HF management | After hospital discharge up to 12 weeks
  A composite number of hospital admissions and emergency department/urgent clinic visits for HF management after admission with ADHF will be documented from electronic medical records (EMR) or as reported by participants.
Participants with symptoms of HF using the Chronic Heart Failure Questionnaire (CHQ-SAS) | Baseline, 6 and 12 weeks
  Participants will complete the CHQ-SAS, a validated questionnaire that assesses patients' perception of their HF and measures the impact of HF symptoms. The CHQ-SAS contains 16 standardized questions that assess dyspnea during daily activities, fatigue, and emotional function. Items are rated on a 7- 7-point Likert scale ranging from 1 to 7.
Quality of life measures using Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline, 6 and 12 weeks
  KCCQ is a disease-specific health status instrument composed of 23 items that quantify physical limitation, symptoms, self-efficacy, social limitation, and quality of life limitation due to HF. Scores range from 0 to 100, with higher scores reflecting better health status. For the KCCQ overall summary score, a small but clinically meaningful change is ≥ 5 points.
Six-minute walk distance (6MWD) | Baseline, 6 and 12 weeks
  Six-minute walk distance measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes. The six-minute walk test serves as a standardized test for functional capacity quantification of HF patients and is predictive of adverse cardiovascular outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Kasra Moazzami, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Grady Health System, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No